CLINICAL TRIAL: NCT03985293
Title: A 16-WEEK, PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO EVALUATE THE EFFICACY AND SAFETY OF TWICE DAILY PF-06882961 ADMINISTRATION IN ADULTS WITH TYPE 2 DIABETES MELLITUS INADEQUATELY CONTROLLED ON METFORMIN OR DIET AND EXERCISE
Brief Title: A 16 Week Study to Evaluate the Efficacy and Safety of PF-06882961 in Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3421005; 2019-000218-12 (EudraCT Number)
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-06882961 2.5 milligrams (mg) (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 10 mg (Experimental)
  Interventions: Drug: PF-06882961
- PF-06882961 40 mg (Experimental): Participants will be titrated up to 2 weeks to reach desired dose level
  Interventions: Drug: PF-06882961
- PF-06882961 80 mg (Experimental): Participants will be titrated up to 4 weeks to reach desired dose level
  Interventions: Drug: PF-06882961
- PF-06882961 120 mg (Experimental): Participants will be titrated up to 6 weeks to reach desired dose level
  Interventions: Drug: PF-06882961

INTERVENTIONS:
Drug: Placebo — 4 matching placebo tablets taken twice a day (BID)
  Arms: Placebo
Drug: PF-06882961 — Participants will be randomized to one of 5 active doses (2.5, 10, 40, 80, or 120 mg), taking 4 tablets twice daily for 16 weeks.
  Arms: PF-06882961 10 mg; PF-06882961 120 mg; PF-06882961 2.5 milligrams (mg); PF-06882961 40 mg; PF-06882961 80 mg

SUMMARY:
This multicenter, randomized, double-blind, placebo controlled, parallel group study is being conducted to provide data on efficacy, safety, tolerability and pharmacokinetics (PK) of multiple dose levels of PF-06882961 in adults with type 2 diabetes mellitus (T2DM) inadequately controlled on metformin and/or diet and exercise. In addition, the study is intended to enable selection of efficacious doses for future clinical development of PF-06882961.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who are treated with metformin and/or diet and exercise
* HbA1c greater than or equal to 7% and less than or equal to 10.5%
* Total body weight >50 kg (110 lb) with BMI 24.5 to 45.4 kg/m^2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* Diagnosis of Type 1 diabetes
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, heart failure, or transient ischemic attack within 6 months of screening
* Any malignancy not considered cured
* Personal or family history of MTC or MEN2, or participants with suspected MTC
* Acute pancreatitis or history of chronic pancreatitis
* Symptomatic gallbladder disease
* Known medical history of active proliferative retinopathy and/or macular edema
* Known medical history of active liver disease, including chronic active hepatitis B or C, or primary biliary cirrhosis
* Known history of HIV
* Supine blood pressure greater than or equal to 160 mmHg (systolic) or greater than or equal to 100 mmHg (diastolic)
* Clinically relevant ECG abnormalities
* Positive urine drug test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (41):
  - Holy Trinity Medical Clinic, Harbor City, California
  - Innovative Clinical Research, Inc., Harbor City, California
  - Long Beach Clinical Trials Services, Inc., Long Beach, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Empire Clinical Research, Pomona, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Incorporated, Tustin, California
  - San Fernando Valley Health Institute, LLC, Van Nuys, California
  - Diablo Clinical Research Incorporated, Walnut Creek, California
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - New Horizon Research Center, Miami, Florida
  - NewPhase Clinical Trials, Corp., Miami Beach, Florida
  - Sunshine Research Center, Inc, Opa-locka, Florida
  - Andres Patron D.O. P.A., Pembroke Pines, Florida
  - Ellipsis Group, Alpharetta, Georgia
  - East Coast Institute for Research, LLC, Macon, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Buynak Clinical Research, Valparaiso, Indiana
  - Viable Research Management LLC, Henderson, Nevada
  - Premier Research, Trenton, New Jersey
  - PharmQuest, Greensboro, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Velocity Clinical Research, Cincinnati, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - Family Medical Associates, Levittown, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Palmetto Primary Care Physicians (physicals only), Summerville, South Carolina
  - Dallas Diabetes Research Center, Dallas, Texas
  - Endocrine Associates, Houston, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Northeast Clinical Research of San Antonio, Live Oak, Texas
  - Sun Research Institute, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Bulgaria (6):
  - MHAT Dobrich AD, Dobrich
  - Medical Center ASKLEPII OOD, Dupnitsa
  - UMHAT Pulmed, Plovdiv
  - Fourth MHAT - Sofia EAD, Sofia
  - MHAT "Doverie" AD, Sofia
  - MC "New rehabilitation center" EOOD, Stara Zagora
- Canada (10):
  - GA Research Associates Ltd., Moncton, New Brunswick
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Manna Research (Toronto), Toronto, Ontario
  - Manna Research (Quebec), Lévis, Quebec
  - Manna Research (Mirabel), Mirabel, Quebec
  - Diex Recherche Quebec Inc., Québec, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Victoriaville Inc., Victoriaville, Quebec
  - Centre de Recherche Saint-Louis, Québec
- Hungary (5):
  - Belinus Orvosi es Szamitastechnikai Bt, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - CRU Hungary Kft., Miskolc
  - Borbanya Praxis Egeszsegugyi KFT, Nyíregyháza
  - Clinfan Kft., Szekszárd
- Poland (6):
  - Zdrowie Osteo-Medic s.c. Lidia i Artur Racewicz, Agnieszka i Jerzy Supronik, Bialystok
  - Medyczne Centrum Diabetologiczno-Endokrynologiczno-Metaboliczne DIAB-ENDO-MET Sp. z o. o., Krakow
  - Prywatny Gabinet Lekarski i Wizyty Lekarskie Jan Ruxer, Lodz
  - MEDICOME Sp. z o.o., Oświęcim
  - KO-MED CENTRA KLINICZNE Sp. z o.o. Ośrodek Badań Klinicznych w Puławach, Puławy
  - Centralny Szpital Kliniczny MSWiA, Warsaw
- Slovakia (7):
  - Metabol KLINIK s.r.o., Bratislava
  - Medispektrum, s.r.o, Bratislava
  - HUMAN-CARE, s.r.o., Košice
  - SchronerMED s.r.o., Moldava nad Bodvou
  - Funkystuff, s.r.o., Nové Zámky
  - DIAB s.r.o., Rožňava
  - MUDr. Jana Rociakova, s.r.o., Žilina
- South Korea (4):
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Samsung Medical Center, Gangnam-Gu, Seoul
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Saxena AR, Frias JP, Brown LS, Gorman DN, Vasas S, Tsamandouras N, Birnbaum MJ. Efficacy and Safety of Oral Small Molecule Glucagon-Like Peptide 1 Receptor Agonist Danuglipron for Glycemic Control Among Patients With Type 2 Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314493. doi: 10.1001/jamanetworkopen.2023.14493. PMID 37213102
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 859 participants were screened in the study, among whom, 412 participants were randomized, and 411 participants were treated with PF-06882961 (Danuglipron)/placebo; 1 participant randomized to the PF-06882961 120 mg BID group was not treated.
Groups:
- Placebo: Placebo matched to PF-06882961 was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up.
- PF-06882961 2.5mg BID: PF-06882961 2.5 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up.
- PF-06882961 10mg BID: PF-06882961 10 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up.
- PF-06882961 40mg BID: PF-06882961 40 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up. Titration was implemented.
- PF-06882961 80mg BID: PF-06882961 80 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up. Titration was implemented.
- PF-06882961 120mg BID: PF-06882961 120 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up. Titration was implemented.
Period: DOUBLE-BLIND TREATMENT
Arm/Group | Placebo | PF-06882961 2.5mg BID | PF-06882961 10mg BID | PF-06882961 40mg BID | PF-06882961 80mg BID | PF-06882961 120mg BID
Started | 66 | 68 | 68 | 71 | 67 | 71
Completed | 57 | 54 | 63 | 57 | 47 | 38
Not Completed | 9 | 14 | 5 | 14 | 20 | 33
Not completed — Adverse Event | 5 | 2 | 3 | 8 | 15 | 24
Not completed — Lost to Follow-up | 1 | 3 | 0 | 3 | 3 | 1
Not completed — No Longer Meets Eligibility Criteria | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 2 | 0 | 1 | 7
Period: FOLLOW-UP
Arm/Group | Placebo | PF-06882961 2.5mg BID | PF-06882961 10mg BID | PF-06882961 40mg BID | PF-06882961 80mg BID | PF-06882961 120mg BID
Started | 57 | 54 | 63 | 57 | 47 | 38
Completed | 57 | 54 | 62 | 57 | 47 | 38
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 412 participants were assigned to treatment, 411 of whom were treated; 1 participant randomized to the PF-06882961 120 mg BID group was not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06882961 2.5mg BID | PF-06882961 10mg BID | PF-06882961 40mg BID | PF-06882961 80mg BID | PF-06882961 120mg BID | Total
Number analyzed (Participants) | 66 | 68 | 68 | 71 | 67 | 71 | 411
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 57.9 (10.27) | 58.9 (9.30) | 58.1 (9.43) | 59.6 (8.58) | 58.4 (9.18) | 58.8 (9.43) | 58.6 (9.33)
Age, Customized [Number; unit: Participants]
  18-44 Years | 6 | 4 | 7 | 2 | 5 | 8 | 32
  45-64 Years | 44 | 43 | 41 | 45 | 42 | 44 | 259
  >=65 Years | 16 | 21 | 20 | 24 | 20 | 19 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 33 | 37 | 32 | 37 | 202
  Male | 33 | 38 | 35 | 34 | 35 | 34 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 22 | 17 | 24 | 23 | 18 | 128
  Not Hispanic or Latino | 42 | 46 | 50 | 47 | 44 | 52 | 281
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 57 | 53 | 58 | 59 | 59 | 343
  Black or African American | 2 | 4 | 10 | 6 | 1 | 4 | 27
  Asian | 5 | 7 | 4 | 6 | 6 | 7 | 35
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Not reported | 1 | 0 | 1 | 1 | 1 | 0 | 4
Age Range [Median (Full Range); unit: Years] | 59.0 [28 to 76] | 59.0 [38 to 74] | 60.0 [38 to 75] | 61.0 [31 to 75] | 58.0 [35 to 75] | 60.0 [40 to 74] | 59.0 [28 to 76]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 16
Description: HbA1c can be used as a diagnostic test for diabetes. The target HbA1c level for people with diabetes is usually less than 7%.
Time Frame: Baseline, Week 16
Population: Overall number of participants analyzed included all participants randomly assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Groups:
- PF-06882961 2.5 BID: PF-06882961 2.5 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up.
- PF-06882961 10 mg BID: PF-06882961 10 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up.
- PF-06882961 40 mg BID: PF-06882961 40 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up. Titration was implemented.
- PF-06882961 80 mg BID: PF-06882961 80 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up. Titration was implemented.
- PF-06882961 120 mg BID: PF-06882961 120 mg was administered orally twice daily (BID) with food for a total of 16 weeks, followed by an approximate 4-week follow-up. Titration was implemented.
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 52 | 52 | 61 | 55 | 46 | 38
Percent | -0.02 [-0.22 to 0.19] | -0.49 [-0.70 to -0.28] | -0.91 [-1.11 to -0.72] | -1.03 [-1.23 to -0.83] | -0.96 [-1.18 to -0.74] | -1.18 [-1.41 to -0.95]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0071, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.47, 90% CI 2-sided [-0.76 to -0.18] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.90, 90% CI 2-sided [-1.18 to -0.62] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -1.01, 90% CI 2-sided [-1.30 to -0.73] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.94, 90% CI 2-sided [-1.24 to -0.65] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -1.16, 90% CI 2-sided [-1.47 to -0.86] — PF-06882961 = Test Placebo = Reference

2. Secondary Outcome: Percentage of Participants Achieving Less Than (<) 7% Glycated Hemoglobin (HbA1c) Levels
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 52 | 52 | 61 | 55 | 46 | 38
Percentage of Participants | 7.7 | 30.8 | 54.1 | 58.2 | 65.2 | 60.5
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 5.11, 90% CI 2-sided [1.84 to 14.18] — The Odds ratio model included multiple imputation. PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 16.85, 90% CI 2-sided [6.18 to 45.93] — The Odds ratio model included multiple imputation. PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 18.79, 90% CI 2-sided [7.03 to 50.21] — The Odds ratio model included multiple imputation. PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 23.97, 90% CI 2-sided [8.66 to 66.39] — The Odds ratio model included multiple imputation. PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 24.46, 90% CI 2-sided [8.72 to 68.57] — The Odds ratio model included multiple imputation. PF-06882961 = Test Placebo = Reference

3. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 2
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 65 | 64 | 67 | 67 | 63 | 69
Percent | -0.09 [-0.17 to -0.01] | -0.18 [-0.26 to -0.09] | -0.31 [-0.39 to -0.23] | -0.29 [-0.37 to -0.21] | -0.33 [-0.41 to -0.24] | -0.35 [-0.43 to -0.28]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.1578, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.09, 90% CI 2-sided [-0.19 to 0.01] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.22, 90% CI 2-sided [-0.32 to -0.12] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.0013, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.20, 90% CI 2-sided [-0.30 to -0.10] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.24, 90% CI 2-sided [-0.34 to -0.14] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.26, 90% CI 2-sided [-0.36 to -0.16] — PF-06882961 = Test Placebo = Reference

4. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 60 | 58 | 68 | 63 | 54 | 60
Percent | -0.08 [-0.19 to 0.04] | -0.38 [-0.50 to -0.26] | -0.51 [-0.62 to -0.39] | -0.63 [-0.74 to -0.52] | -0.58 [-0.70 to -0.46] | -0.64 [-0.75 to -0.53]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0013, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.30, 90% CI 2-sided [-0.46 to -0.15] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.43, 90% CI 2-sided [-0.58 to -0.28] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.55, 90% CI 2-sided [-0.70 to -0.40] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.50, 90% CI 2-sided [-0.66 to -0.35] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.56, 90% CI 2-sided [-0.71 to -0.41] — PF-06882961 = Test Placebo = Reference

5. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 6
Description: as for outcome 1
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 60 | 55 | 66 | 59 | 51 | 52
Percent | -0.07 [-0.21 to 0.07] | -0.47 [-0.61 to -0.34] | -0.71 [-0.84 to -0.57] | -0.84 [-0.97 to -0.71] | -0.79 [-0.93 to -0.65] | -0.84 [-0.98 to -0.71]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.40, 90% CI 2-sided [-0.59 to -0.22] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.64, 90% CI 2-sided [-0.81 to -0.46] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.77, 90% CI 2-sided [-0.95 to -0.59] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.72, 90% CI 2-sided [-0.91 to -0.53] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.77, 90% CI 2-sided [-0.95 to -0.59] — PF-06882961 = Test Placebo = Reference

6. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 56 | 51 | 66 | 58 | 45 | 42
Percent | -0.13 [-0.29 to 0.03] | -0.50 [-0.66 to -0.34] | -0.78 [-0.93 to -0.62] | -0.97 [-1.13 to -0.82] | -0.92 [-1.09 to -0.76] | -1.02 [-1.18 to -0.86]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0054, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.37, 90% CI 2-sided [-0.59 to -0.15] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS Mean = -0.65, 90% CI 2-sided [-0.86 to -0.44] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.84, 90% CI 2-sided [-1.06 to -0.63] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.80, 90% CI 2-sided [-1.02 to -0.57] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.89, 90% CI 2-sided [-1.11 to -0.67] — PF-06882961 = Test Placebo = Reference

7. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 55 | 53 | 63 | 58 | 46 | 38
Percent | -0.09 [-0.28 to 0.10] | -0.53 [-0.72 to -0.34] | -0.88 [-1.06 to -0.70] | -1.06 [-1.25 to -0.88] | -0.91 [-1.12 to -0.71] | -1.11 [-1.32 to -0.91]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0061, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.44, 90% CI 2-sided [-0.71 to -0.18] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.79, 90% CI 2-sided [-1.05 to -0.54] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.98, 90% CI 2-sided [-1.24 to -0.72] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.83, 90% CI 2-sided [-1.10 to -0.56] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -1.03, 90% CI 2-sided [-1.30 to -0.75] — PF-06882961 = Test Placebo = Reference

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 2
Description: The fasting plasma glucose test measures the levels of glucose (sugar) in the blood, with a normal range of 70 milligram per deciliter (mg/dL) to 99 mg/dL.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 65 | 64 | 67 | 68 | 63 | 68
mg/dL | -5.58 [-12.66 to 1.49] | -22.72 [-29.78 to -15.65] | -21.96 [-28.91 to -15.01] | -27.79 [-34.60 to -20.98] | -24.18 [-31.28 to -17.08] | -30.92 [-37.66 to -24.17]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0014, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -17.13, 90% CI 2-sided [-25.94 to -8.33] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.0021, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -16.38, 90% CI 2-sided [-25.08 to -7.67] — Difference in LS Mean
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -22.20, 90% CI 2-sided [-30.88 to -13.53] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -18.59, 90% CI 2-sided [-27.43 to -9.76] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -25.33, 90% CI 2-sided [-34.00 to -16.67] — PF-06882961 = Test Placebo = Reference

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 4
Description: The fasting plasma glucose test measures the levels of glucose (sugar) in the blood, with a normal range of 70 mg/dL to 99 mg/dL.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 60 | 58 | 68 | 62 | 55 | 60
mg/dL | -5.98 [-13.62 to 1.66] | -17.77 [-25.46 to -10.09] | -24.66 [-31.98 to -17.35] | -33.42 [-40.83 to -26.00] | -33.34 [-41.25 to -25.44] | -34.06 [-41.52 to -26.60]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0468, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -11.79, 90% CI 2-sided [-21.55 to -2.04] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.0012, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -18.68, 90% CI 2-sided [-28.12 to -9.25] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -27.44, 90% CI 2-sided [-37.03 to -17.85] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -27.36, 90% CI 2-sided [-37.22 to -17.51] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -28.09, 90% CI 2-sided [-37.72 to -18.45] — PF-06882961 = Test Placebo = Reference

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 6
Description: as for outcome 9
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 60 | 55 | 66 | 60 | 51 | 53
mg/dL | -0.88 [-8.62 to 6.86] | -16.78 [-24.67 to -8.89] | -26.41 [-33.88 to -18.94] | -30.89 [-38.47 to -23.30] | -28.36 [-36.51 to -20.21] | -32.65 [-40.44 to -24.87]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0091, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -15.90, 90% CI 2-sided [-25.90 to -5.90] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -25.53, 90% CI 2-sided [-35.18 to -15.89] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -30.01, 90% CI 2-sided [-39.80 to -20.21] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -27.48, 90% CI 2-sided [-37.63 to -17.33] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -31.77, 90% CI 2-sided [-41.77 to -21.78] — PF-06882961 = Test Placebo = Reference

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 8
Description: as for outcome 9
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 57 | 53 | 64 | 58 | 48 | 42
mg/dL | -9.10 [-16.80 to -1.41] | -12.73 [-20.53 to -4.93] | -26.23 [-33.57 to -18.89] | -29.74 [-37.26 to -22.23] | -33.22 [-41.36 to -25.09] | -34.31 [-42.46 to -26.16]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.5449, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -3.63, 90% CI 2-sided [-13.51 to 6.25] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.0031, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -17.12, 90% CI 2-sided [-26.62 to -7.63] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -20.64, 90% CI 2-sided [-30.31 to -10.96] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -24.12, 90% CI 2-sided [-34.20 to -14.04] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -25.21, 90% CI 2-sided [-35.44 to -14.97] — PF-06882961 = Test Placebo = Reference

12. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 12
Description: as for outcome 9
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 55 | 53 | 63 | 58 | 46 | 37
mg/dL | 1.21 [-7.93 to 10.35] | -6.49 [-15.70 to 2.73] | -22.56 [-31.17 to -13.95] | -32.01 [-40.89 to -23.14] | -30.45 [-40.26 to -20.64] | -32.38 [-42.83 to -21.94]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.2940, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -7.70, 90% CI 2-sided [-19.78 to 4.38] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -23.77, 90% CI 2-sided [-35.37 to -12.17] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -33.23, 90% CI 2-sided [-45.05 to -21.40] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -31.66, 90% CI 2-sided [-44.14 to -19.19] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -33.59, 90% CI 2-sided [-46.67 to -20.51] — PF-06882961 = Test Placebo = Reference

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 16
Description: as for outcome 9
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 52 | 52 | 61 | 56 | 45 | 38
mg/dL | 1.31 [-7.58 to 10.20] | -12.81 [-21.71 to -3.91] | -24.53 [-32.88 to -16.18] | -30.47 [-39.06 to -21.87] | -25.71 [-35.15 to -16.26] | -31.93 [-41.73 to -22.13]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.0464, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -14.12, 90% CI 2-sided [-25.77 to -2.47] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -25.84, 90% CI 2-sided [-37.05 to -14.62] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -31.78, 90% CI 2-sided [-43.20 to -20.35] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -27.02, 90% CI 2-sided [-39.03 to -15.01] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -33.24, 90% CI 2-sided [-45.63 to -20.84] — PF-06882961 = Test Placebo = Reference

14. Secondary Outcome: Change From Baseline in Body Weight at Week 2
Description: Weight was recorded using a calibrated scale (with the same scale used if possible for the duration of the study) reporting weight in kilograms (kg), and accuracy to the nearest 0.1 kg.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 65 | 64 | 68 | 68 | 63 | 69
Kilogram | -0.15 [-0.47 to 0.17] | -0.09 [-0.41 to 0.23] | -0.12 [-0.44 to 0.19] | -0.23 [-0.54 to 0.08] | -0.57 [-0.89 to -0.24] | -0.54 [-0.85 to -0.24]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.8011, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.06, 90% CI 2-sided [-0.33 to 0.44] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.9149, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.02, 90% CI 2-sided [-0.35 to 0.40] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.7216, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.08, 90% CI 2-sided [-0.46 to 0.30] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0758, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.42, 90% CI 2-sided [-0.80 to -0.03] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p = 0.0860, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.40, 90% CI 2-sided [-0.77 to -0.02] — PF-06882961 = Test Placebo = Reference

15. Secondary Outcome: Change From Baseline in Body Weight at Week 4
Description: as for outcome 14
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 61 | 58 | 68 | 63 | 55 | 61
Kilogram | -0.25 [-0.64 to 0.15] | -0.33 [-0.72 to 0.07] | -0.08 [-0.46 to 0.30] | -0.77 [-1.15 to -0.39] | -1.05 [-1.45 to -0.64] | -1.33 [-1.71 to -0.95]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.7898, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.08, 90% CI 2-sided [-0.59 to 0.42] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.5829, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.16, 90% CI 2-sided [-0.33 to 0.66] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.0827, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.52, 90% CI 2-sided [-1.02 to -0.03] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0101, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.80, 90% CI 2-sided [-1.31 to -0.29] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -1.09, 90% CI 2-sided [-1.59 to -0.59] — PF-06882961 = Test Placebo = Reference

16. Secondary Outcome: Change From Baseline in Body Weight at Week 6
Description: as for outcome 14
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 60 | 55 | 66 | 60 | 51 | 53
Kilogram | -0.09 [-0.57 to 0.40] | -0.19 [-0.68 to 0.31] | -0.32 [-0.78 to 0.15] | -0.83 [-1.31 to -0.36] | -1.69 [-2.20 to -1.19] | -2.34 [-2.83 to -1.85]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.7985, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.10, 90% CI 2-sided [-0.75 to 0.55] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.5484, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.23, 90% CI 2-sided [-0.86 to 0.40] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.0541, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.75, 90% CI 2-sided [-1.38 to -0.11] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -1.60, 90% CI 2-sided [-2.26 to -0.95] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -2.25, 90% CI 2-sided [-2.90 to -1.60] — PF-06882961 = Test Placebo = Reference

17. Secondary Outcome: Change From Baseline in Body Weight at Week 8
Description: as for outcome 14
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 57 | 54 | 66 | 58 | 48 | 42
Kilogram | -0.36 [-0.89 to 0.16] | -0.05 [-0.59 to 0.49] | -0.27 [-0.78 to 0.23] | -1.09 [-1.60 to -0.57] | -1.97 [-2.52 to -1.42] | -3.31 [-3.85 to -2.77]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.4692, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.31, 90% CI 2-sided [-0.40 to 1.03] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.8274, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.09, 90% CI 2-sided [-0.60 to 0.78] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.0887, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.72, 90% CI 2-sided [-1.42 to -0.02] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -1.61, 90% CI 2-sided [-2.33 to -0.88] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -2.95, 90% CI 2-sided [-3.67 to -2.22] — PF-06882961 = Test Placebo = Reference

18. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Description: as for outcome 14
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 55 | 53 | 63 | 58 | 46 | 38
Kilogram | -0.24 [-0.85 to 0.38] | -0.09 [-0.72 to 0.53] | -0.00 [-0.59 to 0.58] | -1.05 [-1.65 to -0.44] | -2.52 [-3.17 to -1.87] | -3.81 [-4.46 to -3.16]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.7758, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.15, 90% CI 2-sided [-0.70 to 0.99] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.6367, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.23, 90% CI 2-sided [-0.58 to 1.05] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.1082, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.81, 90% CI 2-sided [-1.63 to 0.02] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -2.28, 90% CI 2-sided [-3.14 to -1.42] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -3.57, 90% CI 2-sided [-4.44 to -2.70] — PF-06882961 = Test Placebo = Reference

19. Secondary Outcome: Change From Baseline in Body Weight at Week 16
Description: as for outcome 14
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Kilogram
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 52 | 53 | 62 | 57 | 46 | 38
Kilogram | -0.43 [-1.12 to 0.25] | 0.02 [-0.68 to 0.72] | -0.06 [-0.71 to 0.60] | -1.16 [-1.84 to -0.49] | -2.48 [-3.20 to -1.75] | -4.60 [-5.34 to -3.86]
Statistical Analysis 1: Comparison: Placebo vs PF-06882961 2.5 BID; Test type: Superiority; p = 0.4325, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.45, 90% CI 2-sided [-0.50 to 1.41] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 2: Comparison: Placebo vs PF-06882961 10 mg BID; Test type: Superiority; p = 0.4978, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = 0.38, 90% CI 2-sided [-0.54 to 1.30] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 3: Comparison: Placebo vs PF-06882961 40 mg BID; Test type: Superiority; p = 0.1970, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -0.73, 90% CI 2-sided [-1.66 to 0.20] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 4: Comparison: Placebo vs PF-06882961 80 mg BID; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -2.04, 90% CI 2-sided [-3.01 to -1.07] — PF-06882961 = Test Placebo = Reference
Statistical Analysis 5: Comparison: Placebo vs PF-06882961 120 mg BID; Test type: Superiority; p < .0001, Mixed Models Analysis; Mixed Model Repeated Measures (MMRM); Difference in LS Mean = -4.17, 90% CI 2-sided [-5.15 to -3.18] — PF-06882961 = Test Placebo = Reference

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (Adverse Events [AEs] and Serious Adverse Events [SAEs])
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Any such events with initial onset or increasing in severity after the first dose of study treatment were counted as treatment-emergent.
Time Frame: Baseline up to Week 21
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 66 | 68 | 68 | 71 | 67 | 71
Participants
  Number of Participants With Treatment Emergent AEs | 32 | 32 | 31 | 42 | 43 | 44
  Number of Participants With Treatment Emergent SAEs | 1 | 1 | 2 | 6 | 2 | 1

21. Secondary Outcome: Number of Participants With Treatment Emergent Clinical Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology (hemoglobin, hematocrit, erythrocytes, reticulocytes, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils, monocytes, activated partial thromboplastin time, prothrombin time, PT/INR, reticulocytes); chemistry (indirect bilirubin, direct bilirubin, protein, albumin, blood urea nitrogen, creatinine, creatine kinase, urate, calcium, sodium, potassium, chloride, bicarbonate, urine urobilinogen); urinalysis (pH, urine glucose, urine ketones, urine protein, urine hemoglobin, nitrites, leukocyte esterase, urine erythrocytes, urine leukocytes, urine hyaline casts, urine bilirubin); lipid panel (low density lipoprotein cholesterol, high density lipoprotein cholesterol).
Time Frame: Baseline Through Week 21
Population: Overall number of participants analyzed included all participants randomly assigned to study treatment and who took at least 1 dose of study treatment and had at least 1 measurement available.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 65 | 68 | 68 | 71 | 67 | 71
Participants | 60 | 57 | 57 | 57 | 60 | 64

22. Secondary Outcome: Number of Participants With Treatment Emergent Vital Signs Abnormalities
Description: Vital signs abnormality criteria: 1) supine systolic blood pressure (SBP) <90 millimeters of mercury (mmHg); 2) supine diastolic blood pressure (DBP) <50 mmHg; 3) supine pulse rate <40 or >120 beats per minute (bpm); 4) change from baseline (increase or decrease) in supine SBP greater than or equal to (>=) 30 mmHg; 5) change from baseline (increase or decrease) in supine DBP >= 20 mmHg.
Time Frame: Baseline through Week 21
Population: Overall number of participants analyzed included all participants randomly assigned to study treatment, took at least 1 dose of study treatment and had at least 1 measurement available.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 65 | 68 | 68 | 71 | 67 | 71
Participants
  Supine SBP <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Supine SBP increase >=30 mmHg | 3 | 4 | 3 | 3 | 0 | 5
  Supine SBP decrease >=30 mmHg | 4 | 4 | 3 | 5 | 5 | 0
  Supine DBP <50 mmHg | 1 | 0 | 0 | 1 | 0 | 1
  Supine DBP increase >=20 mmHg | 1 | 1 | 2 | 3 | 3 | 3
  Supine DBP decrease >=20 mmHg | 3 | 4 | 1 | 3 | 2 | 1
  Supine pulse rate <40 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Treatment Emergent ECG Abnormalities
Description: ECG categorical abnormality criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) greater than or equal to (>=) 300 millisecond (msec), b) >=25% increase when baseline is > 200 msec or >=50% increase when baseline is less than or equal to (<=) 200 msec.
  2. QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) >=140 msec, b) >=50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and <=480 msec, b) >480 msec and <=500 msec, c) >500 msec, d) >30 msec and <=60 msec increase from baseline, e) >60 msec increase from baseline.
Time Frame: Baseline Through Week 21
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 2.5 BID | PF-06882961 10 mg BID | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 65 | 68 | 68 | 71 | 67 | 71
Participants
  PR interval ≥300 msec: number analyzed (Participants) | 65 | 67 | 68 | 71 | 67 | 71
  PR interval ≥300 msec | 0 | 0 | 0 | 0 | 0 | 1
  %Change in PR interval ≥25/50%: number analyzed (Participants) | 65 | 67 | 68 | 71 | 67 | 71
  %Change in PR interval ≥25/50% | 3 | 0 | 0 | 0 | 1 | 0
  QRS interval ≥140 msec | 1 | 1 | 0 | 0 | 0 | 0
  %Change in QRS interval ≥50% | 1 | 1 | 0 | 0 | 0 | 0
  QTcF interval >450 and ≤480 msec | 2 | 3 | 2 | 1 | 3 | 4
  QTcF interval >480 and ≤500 msec | 0 | 0 | 0 | 0 | 0 | 1
  QTcF interval >500 msec | 0 | 0 | 0 | 0 | 0 | 0
  Change in QTcF interval >30 and ≤60 msec | 2 | 3 | 2 | 6 | 3 | 6
  Change in QTcF interval >60 msec | 0 | 0 | 1 | 1 | 0 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 21
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Placebo | PF-06882961 2.5mg BID | PF-06882961 10mg BID | PF-06882961 40mg BID | PF-06882961 80mg BID | PF-06882961 120mg BID
All-Cause Mortality (participants affected / at risk) | 0/66 | 1/68 | 0/68 | 2/71 | 0/67 | 0/71
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/68 | 2/68 | 6/71 | 2/67 | 1/71
Other Adverse Events (participants affected / at risk) | 15/66 | 21/68 | 17/68 | 33/71 | 40/67 | 35/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | PF-06882961 2.5mg BID (N=68) | PF-06882961 10mg BID (N=68) | PF-06882961 40mg BID (N=71) | PF-06882961 80mg BID (N=67) | PF-06882961 120mg BID (N=71)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=66) | PF-06882961 2.5mg BID (N=68) | PF-06882961 10mg BID (N=68) | PF-06882961 40mg BID (N=71) | PF-06882961 80mg BID (N=67) | PF-06882961 120mg BID (N=71)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 4 | 8 | 12 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 3 | 2 | 9 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 4 | 5
Nausea (Gastrointestinal disorders) | 2 | 5 | 5 | 11 | 22 | 23
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 11 | 18
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 5 | 3 | 1
SARS-CoV-2 test positive (Investigations) | 2 | 4 | 3 | 2 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 2 | 1 | 0 | 4 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 6 | 3
Dizziness (Nervous system disorders) | 1 | 1 | 4 | 3 | 1 | 5
Headache (Nervous system disorders) | 4 | 4 | 1 | 5 | 2 | 7
Hypertension (Vascular disorders) | 0 | 1 | 3 | 1 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT03985293/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT03985293/SAP_001.pdf